CLINICAL TRIAL: NCT04298463
Title: Retrospective Effectiveness Study of Dalbavancin and Other Standard of Care of the Same Class (i.v. Lipo and Glyco-peptides) in Patients With ABSSSI
Brief Title: Retrospective Effectiveness Study of Dalbavancin and Other Standard of Care of the Same Class in Patients With ABSSSI
Acronym: REDS
Status: Completed | Type: Observational
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Hippocrates Research (Other)
Responsible Party: Sponsor
Other Study IDs: 146(A)PO18530
Record Dates: First submitted 2020-02-10; First posted 2020-03-06 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Acute Bacterial Skin and Skin Structure Infection
Keywords: ABSSSI; skin infections; lipoglycopeptide,; Gram-positive bacteria
MeSH Terms: conditions — Cellulitis | interventions — dalbavancin; Vancomycin; Teicoplanin; Daptomycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COHORT A: dalbavancin: Patients hospitalized for at teast two days affected by ABSSSI and treated with dalbavancin.
  Interventions: Drug: Xydalba
- COHORT B: lipo and glyco-peptid drugs: Patients hospitalized for at teast two days affected by ABSSSI and treated with vancomycin, teicoplanin or daptomycin.
  Interventions: Drug: vancomycin, teicoplanin or daptomycin

INTERVENTIONS:
Drug: Xydalba — Drugs were administered i.v.
  Groups: COHORT A: dalbavancin
Drug: vancomycin, teicoplanin or daptomycin — Drugs were administered i.v.
  Groups: COHORT B: lipo and glyco-peptid drugs

SUMMARY:
The aim of this study is to collect the data on the effectiveness of dalbavancin in terms of save of hospitalization days on patients treated between June 2017 and June 2019 in two countries (Italy and Greece) vs the other Standards of care of the same class (SoC; i.v. lipo and glycopeptides) in a real-life context.

Time to discharge from the start of therapy for ABSSSI in the hospital context will be assessed and all relevant data available on patient management, clinical, microbiological and safety outcomes during hospitalization and in the follow-up visits up to 30 days from discharge will be collected and evaluated.

DETAILED DESCRIPTION:
Acute bacterial skin and skin structure infections (ABSSSI), formally referred to as complicated skin and soft tissue infections, include infections such as cellulitis/erysipelas, wound infection, and major cutaneous abscess and have a minimum lesion surface area of approximately 75 cm2. The regulatory definitions of major abscess, cellulitis, and wound infection may not align with practice-based criteria. Common bacterial pathogens causing ABSSSI are Streptococcus pyogenes and Staphylococcus aureus including Methicillin-Resistant Staphylococcus Aureus (MRSA). Less common causes include other Streptococcus species, Enterococcus faecalis, or Gram-negative bacteria.

Increasing dramatically in incidence, a challenging medical problem associated with high direct and indirect costs has been highlighted for both the medical system and society.

Over the last decade, there was a witnessed a dramatic increase in the incidence of community acquired skin infections, an increasing proportion of which are a consequence of MRSA, reinforcing the need for new and effective antibacterial therapies in this disease.

In this context, research has been promoted to develop new antibiotics capable to fight MRSA, the most common multi-drug-resistant Gram+ bacterium in Europe, and to overcome the limitations of the most widely used antibiotics, such as vancomycin, teicoplanin, and β- lactams. These new antibiotics (lipoglycopeptides and new oxazolidinones) have innovative characteristics that make them interesting for the specific treatment of ABSSSIs. Dalbavancin is one of these new antibiotics. Dalbavancin is a lipoglycopeptide with activity against Grampositive organisms, including MRSA, through interference with bacterial cell wall formation by preventing cross-linking of peptidoglycans. Dalbavancin has a distinctive pharmacokinetic profile, with a terminal half-life of 14.4 days, which allows for infrequent or even single intravenous dosing.

This new long-acting antibiotic represents a potential opportunity for early discharge. This approach could profoundly modify the management of these infections by reducing or in some cases eliminating hospitalization costs and risks.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥ of 18 years old
2. Patients hospitalized for at least 2 days with evidence of primary diagnosis of ABSSSI of International Classification of Diseases (ICD) 9: - 681.XX (cellulitis and abscess of finger and toe) -682.XX (other cellulitis and abscess) - 958.3X (post-traumatic wound infection not elsewhere classified) - 998.5X (postoperative infection not elsewhere classified); and corresponding code for ICD 10; and/or Diagnosis-related group (DRG) 277; 278; 418 (for Italy), for cellulitis/erysipelas, wound infection, major cutaneous abscess.
3. Patients treated with dalbavancin or other SoC of the same or similar class (i.v. lipo and glycopeptides: teicoplanin, vancomycin, daptomycin) according to summary of product characteristics (SmPC).
4. Patients treated with or without other chemotherapy to cover Gram- bacteria or fungals.
5. Patients who gave their consent for personal data processing according to the local regulation.

Exclusion Criteria:

1. Patients with infected wound or ulcer (neoplastic, inflammatory and autoimmune ulcers), animal bite
2. Patients with ulcer not colonized, discolored, odorous, pressure ulcer grade I, II, III, or IV (according to NPUAP classification - Appendix A)
3. Patients with arteriopathies
4. Patients presenting or who have presented in the last 30 days before the hospitalization the following infections:

   * diabetic foot infection (ICD9= 707.15; 249.8)
   * suspected or confirmed osteomyelitis (ICD9= 730.xx)
   * suspected or confirmed septic arthritis (ICD9= 711.00)
   * infective endocarditis (ICD9=421.0)
   * meningitis (ICD9=322.xx)
   * joint infection (ICD9= 711.00)
   * necrotizing fasciitis (ICD9=728.86)
   * gangrene (ICD9=785.4)
   * prosthetic joint infection or prosthetic implant/device infection (ICD9=996.66)
5. Patient with history of neutropenia or in treatment with immunosuppressants in the last six months before the hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients hospitalized for at least 2 days with evidence of primary diagnosis of ABSSSI and treated with dalbavancin or other SoC of similar class (i.v lipo and glycopeptides vancomycin, teicoplanin or daptomycin).
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
Time of discharge from any ward of the hospital, | From baseline to discharge, an average of 4 weeks
  Time of discharge is calculated as the time elapsed from the beginning of antibiotic therapy (baseline) until discharge.

SECONDARY OUTCOMES:
Evaluation of the recorded signs and symptoms | From the hospital admission until 30 days from discharge
  Evaluation of local signs of inflammation.
Microbiological evaluation | From the hospital admission until 30 days from discharge
  Eradication of the Gram Positive pathogens identified at baseline (MIC assessment)
Long-term follow-up | 90 days from discharge
  Assessment for recurrence of ABSSSI.

CONTACTS AND LOCATIONS:
Locations (16):
- Greece (4):
  - University Hospital of Alexandroupolis, Alexandroupoli
  - Attikon University Hospital, Rimini 1, Chaidari, 124 62, Athens
  - University Hospital of Heraklion, Heraklion
  - University General Hospital of Thessaloniki AHEPA /, Thessaloniki
- Italy (12):
  - AO Sant'Orsola Malpighi Unità Operativa di Malattie Infettive, Bologna
  - Azienda Ospedaliera per l'Emergenza Cannizzaro Unità Operativa Complessa di Malattie Infettive, Catania
  - A.O.U. Careggi SOD Malattie Infettive e Tropicali, Florence
  - Ospedale Policlinico San Martino - IRCCS Genova Clinica Malattie Infettive, Genova
  - ASST MANTOVA Ospedale Carlo Poma di Mantova S.C. Malattie Infettive, Mantova
  - A.S.S.T. GRANDE OSPEDALE METROPOLITANO NIGUARDA S.C. Malattie Infettive Dipartimento Medico Polispecialistico, Milan
  - AOU Federico II di Napoli Dipartimento di Medicina clinica e Chirurgia UOC Malattie Infettive, Napoli
  - Azienda Ospedaliera di Padova U.O.C. Malattie Infettive e Tropicali, Padua
  - Ospedale S. Maria della Misericordia Clinica Malattie Infettive Dipartimento di Medicina, Università Studi di Perugia, Perugia
  - A.O.U. Pisana Stabilimento di Cisanello U.O Malattie Infettive, Pisa
  - A.O.R. San Carlo Struttura Interaziendale Complessa di Malattie Infettive, Potenza
  - AOU Città della Salute e Scienza - Presidio Molinette SC Malattie Infettive, Torino